CLINICAL TRIAL: NCT02765477
Title: Paced Electrocardiogram Requiring Fast Emergent Coronary Therapy (PERFECT) Study
Acronym: PERFECT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hennepin County Medical Center, Minneapolis (Other)
Responsible Party: Principal Investigator, Stephen W. Smith, Faculty Emergency Physician, Professor of Emergency Medicine, Hennepin County Medical Center, Minneapolis
Other Study IDs: HSR 15-4101
Record Dates: First submitted 2016-04-22; First posted 2016-05-06 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute myocardial infarction; ST Elevation Myocardial Infarction; Acute Coronary Occlusion; Electrocardiogram; Ventricular Paced Rhythm; Modified Sgarbossa Criteria
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Angiogram Cohort w Acute Coronary Occlusion: Inclusion Criteria: Angiogram Cohort. Patients who present 1) directly through the study site Emergency Department (ED) OR 2) as a transfer or referral patient from the ED of another institution OR 3) as a direct admission to the study site's Catheterization Laboratory by an ambulance service, who also met the following criteria: 1.Underwent urgent or emergent coronary angiography during the index presentation for suspected ischemic symptoms (including but not limited to chest pain [CP] and/or shortness of breath [SOB]) AND 2. Had a VPR ECG recorded during the index presentation prior to the angiogram AND 3. Had sufficient troponins to rule in or rule out acute myocardial injury, per the study site's institutional protocol. From this Angiogram Cohort, a group of patients will be identified who had angiographic evidence of ACO, defined as an acute lesion with TIMI flow 0 or 1 when evaluated by an experienced study-site adjudicator.
- Non-ACO Angiogram Cohort: Inclusion Criteria: Angiogram Cohort. Each study site will first identify adult patients (age 18 years or older) who presented to the study site 1) directly through the study site ED OR 2) as a transfer or referral patient from the ED of another institution OR 3) as a direct admission to the study site's Catheterization Laboratory by an ambulance service, who also met the following criteria: 1. Underwent coronary angiography during the index presentation for suspected ischemic symptoms (including but not limited to CP and/or SOB AND 2. Had a VPR ECG recorded during the index presentation prior to the angiogram AND 3. Had sufficient troponins to rule in or rule out acute myocardial injury, per the study site's institutional protocol. From this Angiogram Cohort, those who had TIMI-2 or greater flow will be identified for several research questions.
- Random ED Sample w Paced Rhythm but No AMI: Each site will select a random sample of all adult patients who present to the ED (or by ambulance directly to the Catheterization Lab) with suspected ischemic symptoms and a VPR ECG.
  Each study site will randomly select 5 unique encounters for every one 1 ACO subject identified by the site. If a study site identifies no ACO subjects, they will randomly select 30 unique encounters.
  Study subjects who are included as subjects in the Angiogram Cohort (data set #1, above) and who are also selected as part of the random sample (data set #2) will be identified in REDCap as subjects for analysis in both groups, but their data will be submitted only once.
  The primary control group selected from this search will be all patients in this group who do not meet criteria for acute myocardial injury, as defined by 1) all troponins below the 99th percentile or 2) Peak troponin < 3x the upper limit of normal AND no rise and/or fall of > 30%.
- ED Patients w Paced Rhythm Without AMI excluded: Each site will select a random sample of all adult patients who present to the ED (or by ambulance directly to the Catheterization Lab) with suspected ischemic symptoms and a VPR ECG.
  Each study site will randomly 5 unique encounters for every 1 ACO subject identified by the site. If a study site identifies no ACO subjects, they will randomly select 30 unique encounters.
  Study subjects who are included as subjects in the Angiogram Cohort (data set #1, above) and who are also selected as part of the random sample (data set #2) will be identified in REDCap as subjects for analysis in both groups, but their data will be submitted only once.
  The secondary control group will include patients in this group in whom Acute MI cannot be excluded because they either have at least 1 troponin > 3x the upper limit of normal or they have at least 1 troponin between 1x and 3x the ULN AND have a rise and/or fall of at least 30%.

SUMMARY:
The number of patients with cardiovascular implantable electronic devices (CIED), including ventricular pacemakers, continues to increase. However, there are no accurate electrocardiographic (ECG) criteria to diagnose acute myocardial infarction (AMI), even if due to acute coronary occlusion (ACO), with a ventricular pacemaker in situ. In this retrospective, multicenter, case-control study the investigators will examine ECG criteria to diagnose ACO in patients with ventricular paced rhythms. During this process, the investigators will also create a database from which investigators will be able to answer multiple additional questions on this population of patients.

DETAILED DESCRIPTION:
BACKGROUND Diagnosis and management of ACO (the anatomic substrate for ST-elevation myocardial infarction) is time sensitive. Diagnosis necessitates emergent reperfusion therapy. An important predictor of death from ACO includes time to reperfusion.1 Delays in reperfusion therapy, including primary percutaneous coronary intervention (PCI) or fibrinolysis, are associated with worse 30-day and 1-year mortality. American Heart Association (AHA) guidelines for treatment of ACO recommend that the first medical contact to device time be less than 120 minutes in patients who have no contraindications to treatment.2 Though cardiac biomarkers are helpful in making the diagnosis in uncertain cases, the time sensitive nature of intervention for ACO precludes their use to direct emergent reperfusion therapy. Furthermore, biomarkers do not diagnose ACO but rather any AMI, including those without occlusion that do not need emergent intervention.

The "traditional" ECG diagnosis of ACO, which includes ST-elevation cutoffs based upon age and sex, excludes patients with ventricular paced rhythm (VPR).3 The small field of research on the topic of ACO in VPR has extrapolated and analyzed data from patients with left bundle branch block (LBBB). That is because VPR with right ventricular pacing and LBBB both result in depolarization from right to left through myocardium (not through conducting fibers) and thus result in similar ECG findings (e.g. wide QRS, delayed onset of depolarization, and abnormal repolarization with "discordant" [in the opposite direction of the QRS] T-waves and ST-segment deviation). In the presence of known LBBB, AHA guidelines recommend using the Sgarbossa criteria to make the diagnosis of ACO.4 Sgarbossa et al. proposed requiring at least 3 points from the following criteria for the diagnosis of acute myocardial infarction in the presence of LBBB: (1) concordant ST-segment elevation of 1 mm (0.1 mV) in at least 1 lead (5 points), (2) concordant ST-segment depression of at least 1 mm in leads V1 to V3 (3 points), or (3) excessively discordant ST-segment elevation, defined as greater than or equal to 5 mm of ST-segment elevation when the QRS complex is negative (2 points). There have been only a handful of evaluations of Sgarbossa's criteria in VPR, with variable methodologies and patient populations; sensitivities in the studies ranged from 10-53% and specificities ranged from 84-99%.5,6 Neither study used angiographic endpoints, but only used biomarker definitions of AMI; one study used a very flawed biomarker definition with no adjudication. Thus, the number of occlusions is entirely unknown and probably very small.

For LBBB, Smith et al. derived and validated a "modified Sgarbossa rule" in which they replaced Sgarbossa's third criterion (excessively discordant ST elevation as defined by 5 mm) with a proportion-based criterion (defined by > 25% of the previous S-wave) (see Table 1). This rule resulted in much higher sensitivity and accuracy for diagnosis of ACO than the original Sgarbossa.7,8

Table 1: MODIFIED SGARBOSSA CRITERIA

1. ST-segment elevation >= 1 mm and concordant with the QRS in any lead
2. ST-segment depression >= 1 mm and concordant with the QRS in any of leads V1- V3
3. Proportionally excessive discordant ST-segment elevation in at least one lead, as defined by ST/S (</= -0.25) with at least 1 mm of STE

The modified Sgarbossa criteria have never been evaluated in patients with VPR and very few additional criteria have ever been evaluated. To our knowledge, no criteria have been evaluated using an angiographic outcome, the only outcome relevant to guiding emergency reperfusion therapy. The primary purpose of this study will be to investigate the diagnostic performance of selected ECG criteria for the diagnosis of ACO in VPR. Through the process of answering this question, a database will be formed to answer multiple additional questions on this patient population that is underrepresented in clinical trials.

STUDY DESIGN The primary analysis will be designed as a multicenter, retrospective case-control study. Additionally, data will be collected to create a database of de-identified patient information that will allow researchers to investigate numerous additional questions.

Study sites will include Hennepin County Medical Center (HCMC, the lead site) and academic and community centers (study sites) located internationally. Because AMI was redefined in 2007 by a rise and/or fall of troponin, with at least one value above the 99% reference value,9 our study will only include subjects that presented from January 1, 2008 through December 31, 2015.

ELIGIBILITY:
Inclusion Criteria:

* 18 year old at least, ischemic symptoms (e.g., chest pain, shortness of breath, etc.), ventricular paced rhythm on the Electrocardiogram (ECG).

Exclusion Criteria:

* Exclusion from Primary Analysis:

  1. Extreme tachycardia (heart rate > 130 bpm) at the time of presentation
  2. Severe hypertension (diastolic blood pressure > 120 mmHg) at the time of presentation
  3. Respiratory failure (defined as need for positive pressure ventilation) due to pulmonary edema at the time of presentation.
  4. Hyperkalemia (serum potassium > 5.5 mEq/L) at the time of presentation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: I. Adults who presented either 1) directly through the Emergency Department (ED), 2) as a transfer or referral patient, or 3) as a direct ambulance admission to the Catheterization Laboratory, who also:
  1. Underwent urgent or emergent coronary angiography during the index presentation for suspected ischemic symptoms, and
  2. Had a ventricular paced rhythm (VPR) on the ECG
  3. Had sufficient troponins to rule in or rule out acute myocardial injury, per the study site's institutional protocol.
  II. Next, each study site will identify all adult ED patients with a VPR ECG recorded during the index presentation who presented with suspected ischemic symptoms. Simple random selection will be used to identify subjects from this population. There may be overlap between this group and the angiogram group above and this will be considered at the data analysis stage (see Procedures Manual for more detail).
  The first group will not be a probability sample, but the second group will be.
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-04 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and Specificity of Modified Sgarbossa Criteria for Diagnosis of Acute Coronary Occlusion in the Setting of Ventricular Paced Rhythm in Patients with Potential Ischemic Symptoms | 7 days

SECONDARY OUTCOMES:
Sensitivity and Specificity of the modified Sgarbossa criteria with criterion #2 extended from electrocardiogram leads V1-V3 to leads V1-V6 | 7 days
Performance characteristics of the modified Sgarbossa criteria using a maximum ST/S ratio of -0.20, and of -0.30, instead of -0.25 | 7 days
Performance characteristics of absolute ECG millimeter measurements of ST discordance (including both discordant ST elevation and ST depression), using various ratio cutoffs (e.g. -0.2, -0.25, -0.3). | 7 days
Performance characteristics of 0.5 mm (vs. 1 mm) concordant ST-deviation. | 7 days
Performance characteristics of non-concave ST-morphology | 7 days
Mean QRS amplitude of occlusion vs. no occlusion groups. Plot receiver-operator curve for QRS amplitude | 7 days
Find mean T-wave amplitude in occlusion vs. no occlusion groups. Plot ROC curves for T/QRS ratio between groups. | 7 days
Mean QTc, JTc, and TpTe in occlusion vs no occlusion groups, and plot ROC curves for QTc, JTc, and TpTe | 7 days
Multivariate regression model including measurements of concordant and discordant ST elevation or depression, and of QRS amplitude, all in millimeters, and of repolarization time, in milliseconds. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth W Dodd, M.D., Study Chair — Hennepin County Medical Center, Minneapolis, MN; Stephen W Smith, M.D., Principal Investigator — Hennepin County Medical Center, Minneapolis, MN; Deborah L Zvosec, Ph.D., Study Director — Hennepin Healthcare Research Institute; Rehan Karim, MBBS, Study Chair — Hennepin County Medical Center, Minneapolis, MN; Louise Cullen, MD, Study Chair — Royal Brisbane and Women's Hospital; Richard Body, MD, PhD, Study Chair — The University of Manchester
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] O'Gara PT, Kushner FG, Ascheim DD, Casey DE Jr, Chung MK, de Lemos JA, Ettinger SM, Fang JC, Fesmire FM, Franklin BA, Granger CB, Krumholz HM, Linderbaum JA, Morrow DA, Newby LK, Ornato JP, Ou N, Radford MJ, Tamis-Holland JE, Tommaso CL, Tracy CM, Woo YJ, Zhao DX. 2013 ACCF/AHA guideline for the management of ST-elevation myocardial infarction: a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines. J Am Coll Cardiol. 2013 Jan 29;61(4):e78-e140. doi: 10.1016/j.jacc.2012.11.019. Epub 2012 Dec 17. No abstract available. PMID 23256914
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Writing Group on the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Thygesen K, Alpert JS, White HD, Jaffe AS, Katus HA, Apple FS, Lindahl B, Morrow DA, Chaitman BA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S; ESC Committee for Practice Guidelines (CPG). Third universal definition of myocardial infarction. Eur Heart J. 2012 Oct;33(20):2551-67. doi: 10.1093/eurheartj/ehs184. Epub 2012 Aug 24. No abstract available. PMID 22922414
- [Background] Sgarbossa EB. Recent advances in the electrocardiographic diagnosis of myocardial infarction: left bundle branch block and pacing. Pacing Clin Electrophysiol. 1996 Sep;19(9):1370-9. doi: 10.1111/j.1540-8159.1996.tb04217.x. No abstract available. PMID 8880802
- [Background] Jaffe AS. Third universal definition of myocardial infarction. Clin Biochem. 2013 Jan;46(1-2):1-4. doi: 10.1016/j.clinbiochem.2012.10.036. Epub 2012 Nov 2. No abstract available. PMID 23127386
- [Result] Nielsen PH, Terkelsen CJ, Nielsen TT, Thuesen L, Krusell LR, Thayssen P, Kelbaek H, Abildgaard U, Villadsen AB, Andersen HR, Maeng M; Danami-2 Investigators. System delay and timing of intervention in acute myocardial infarction (from the Danish Acute Myocardial Infarction-2 [DANAMI-2] trial). Am J Cardiol. 2011 Sep 15;108(6):776-81. doi: 10.1016/j.amjcard.2011.05.007. Epub 2011 Jul 15. PMID 21757183
- [Result] Sgarbossa EB, Pinski SL, Barbagelata A, Underwood DA, Gates KB, Topol EJ, Califf RM, Wagner GS. Electrocardiographic diagnosis of evolving acute myocardial infarction in the presence of left bundle-branch block. GUSTO-1 (Global Utilization of Streptokinase and Tissue Plasminogen Activator for Occluded Coronary Arteries) Investigators. N Engl J Med. 1996 Feb 22;334(8):481-7. doi: 10.1056/NEJM199602223340801. PMID 8559200
- [Result] Maloy KR, Bhat R, Davis J, Reed K, Morrissey R. Sgarbossa Criteria are Highly Specific for Acute Myocardial Infarction with Pacemakers. West J Emerg Med. 2010 Sep;11(4):354-7. PMID 21079708
- [Result] Meyers HP, Limkakeng AT Jr, Jaffa EJ, Patel A, Theiling BJ, Rezaie SR, Stewart T, Zhuang C, Pera VK, Smith SW. Validation of the modified Sgarbossa criteria for acute coronary occlusion in the setting of left bundle branch block: A retrospective case-control study. Am Heart J. 2015 Dec;170(6):1255-64. doi: 10.1016/j.ahj.2015.09.005. Epub 2015 Sep 24. PMID 26678648
- [Result] Smith SW, Dodd KW, Henry TD, Dvorak DM, Pearce LA. Diagnosis of ST-elevation myocardial infarction in the presence of left bundle branch block with the ST-elevation to S-wave ratio in a modified Sgarbossa rule. Ann Emerg Med. 2012 Dec;60(6):766-76. doi: 10.1016/j.annemergmed.2012.07.119. Epub 2012 Aug 31. PMID 22939607